CLINICAL TRIAL: NCT03552861
Title: Standardization and Optimization of TMS Protocols for the Treatment of Early and Mild-to-late Stage Parkinson's Disease With Depression or Cognitive Impairment
Brief Title: Standardization and Optimization of TMS Protocols for the Treatment of PD With Depression or Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDREC2017083H（R1）
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-07

CONDITIONS: TMS Protocols in the Treatment of PD
Keywords: Parkinson's disease; rTMS; Dorsal prefrontal cortex; Depression; Cognitive impairment
MeSH Terms: conditions — Parkinson Disease; Depression; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- left and right DLPFC active treatment (Active Comparator): Intervention: repetitive transcranial stimulation (rTMS) Each patient will be given 5 treatment sessions per week for 2 weeks (a total of 10 sessions).In each rTMS conditioning session,1200 pulses of stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left and rigt DLPFC.Each session is 45 minutes long and will be consisted of 10Hz stimulation trains (active) over the left DLPFC and 1Hz over the right DLPFC，Interval of 5 minutes each side.During rTMS blocks, the coil will be oriented tangential to the surface.
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)
- left DLPFC active and right DLPFC sham treatment group (Active Comparator): Each patient will be given 5 treatment sessions per week for 2 weeks (a total of 10 sessions).In each rTMS conditioning session,1200 pulses of stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left and rigt DLPFC.Each session is 45 minutes long and will be consisted of 10Hz stimulation trains (active) over the left DLPFC and 1Hz over the right DLPFC，Interval of 5 minutes each side.During rTMS blocks, the coil will be oriented tangential to the surface. For sham control rTMS blocks, the coil will be oriented 90◦ away from the scalp so that no pulses perturbed underlying neural tissue.
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)
- left DLPFC sham and right DLPFC active treatment group (Active Comparator): Each patient will be given 5 treatment sessions per week for 2 weeks (a total of 10 sessions).In each rTMS conditioning session,1200 pulses of stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left and rigt DLPFC.Each session is 45 minutes long and will be consisted of 10Hz stimulation trains (active) over the left DLPFC and 1Hz over the right DLPFC，Interval of 5 minutes each side.During rTMS blocks, the coil will be oriented tangential to the surface. For sham control rTMS blocks, the coil will be oriented 90◦ away from the scalp so that no pulses perturbed underlying neural tissue.
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)
- left DLPFC sham and right DLPFC sham treatment group (Sham Comparator): Each patient will be given 5 treatment sessions per week for 2 weeks (a total of 10 sessions).In each rTMS conditioning session,1200 pulses of stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left and rigt DLPFC.Each session is 45 minutes long and will be consisted of 10Hz stimulation trains (active) over the left DLPFC and 1Hz over the right DLPFC，Interval of 5 minutes each side.During rTMS blocks,the coil will be oriented 90◦ away from the scalp so that no pulses perturbed underlying neural tissue.
  Interventions: Device: repetitive transcranial magnetic stimulation(rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation(rTMS) — Each patient will be given 5 treatment sessions per week for 2 weeks (a total of 10 sessions).In each rTMS conditioning session,1200 pulses of stimuli at an intensity of 100% rest motor threshold (RMT) will give over the left and rigt DLPFC.Each session is 45 minutes long and will be consisted of 10Hz stimulation trains (active) over the left DLPFC and 1Hz over the right DLPFC，Interval of 5 minutes each side.During rTMS blocks, the coil will be oriented tangential to the surface. For sham control rTMS blocks, the coil will be oriented 90◦ away from the scalp so that no pulses perturbed underlying neural tissue.

SUMMARY:
The goal of this study is to determine whether transcranial magnetic stimulation (TMS) is an effective treatment in Parkinson's disease patients with depression or cognitive impairment. The study consists of seven total visits to all. Compensation will be provided for each visit.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation(TMS) is a valuable non-invasive brain stimulation tool for interventional neurophysiology applications, which generate local current and modulates brain activity in a specific, cortico-subcortical network. Repetitive TMS (rTMS) is developed as it is safe and well-tolerated. The left dorsolateral prefrontal cortex (DLPFC) high-frequency rTMS treatment has been proved effective for depression by many clinical studies,as well as the low-frequency rTMS over the right DLPFC. In Europe, guidelines on the therapeutic use of rTMS was published in 2014, in which they pointed out that high-frequency rTMS over left DLPFC could be used as therapeutic method for dPD, with a B-level recommendation. Among several small and pilot studies of rTMS in PD patients, rTMS over either the motor cortex or DLPFC has been reported to show beneficial effects on cognitive impairment with no serious adverse events.However, the relative effectiveness of rTMS over left or right prefrontal, or both regions on both depression and cognitive impairment symptoms, has yet to be established in PD patients.

The investigators propose to conduct a ten-center, blinded, sham-controlled, randomized, parallel-group study of fixed-dose, high-frequency and/or low-frequency rTMS in 252 PD patients who are experiencing depressive symptoms or cognitive impairment. Subjects will be randomized to receive rTMS over right and left DLPFC, both or neither active/sham rTMS. Subjects will receive rTMS for 45 minutes treatment over a 2-week period, all subjects will undergo a comprehensive assessment of mood, cognition, motor and quality of life before and after the last rTMS treatment, and after 2,4 and 12 weeks post-treatment. This study directly addresses the expansion of rTMS as an alternative treatment for depression and cognitive impairment in the PD population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 80 years old, male or female
2. Subjects with idiopathic PD (according to Movement Disorder Society Clinical Diagnostic Criteria，both clinically established PD and clinically probable PD)
3. Subjects fulfilling the criteria of the Diagnostic and Statistical Manual of Mental Disorders, 4th edition(DSM-IV)
4. Did not use antidepressant(s) for a minimum of 2 months
5. Untreated or had stabilized doses of anti-Parkinson's disease medication for > 28 days, and maintain this dose during treatment
6. Subjects or their legal representatives could follow the research plan, visit plan
7. Subjects or their legal guardians agree to participate in the trial and signs informed consent

Exclusion Criteria:

1. Subjects with Parkinson's plus syndrome(PPS) or Secondary Parkinson Disease caused by vascular factors, toxins, and drugs
2. Subjects with persistent head tremor
3. Subjects with dementia
4. Subjects with suicidal tendency and psychotic symptoms
5. Subjects with consciousness, history of stroke, severe neurological/psychiatric disorders such as transient ischemic attack within 1 year prior to screening (Visit 1), or other severe organic diseases
6. Accepted deep brain stimulation(DBS) or other invasive brain surgery previously
7. Subjects with contraindications for repetitive transcranial magnetic stimulation(rTMS), such as history of epileptic seizures, pregnant, implantation of pacemaker or other metal implants in the body, intracranial hypertension, severe hemorrhagic tendency, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale（HAMD） | 3 months
  The Hamilton Depression Rating Scale (HAMD) is a 24-item interviewer administered structure questionaire designed to assess symptoms of depression. Items are scored with a range of 0-4, though 11 of the items are scored between 0 and 2. A total score is then calculated of all items which can range from 0 to 74. A higher score is indicative of more depressive symptoms, and a lower score post-tx is indicative of better outcome.
Beck Depression Inventory（BDI） | 3 months
  The Beck Depression Inventory (BDI) is a 21-item self-report questionaire that measures depressive symptoms. Each item is scored on a scale of 0-3, and items are summated to yield a total score. A higher score is indicative of greater symptoms of depression. Total scores may range between 0 and 63. A score greater than or equal of 14 is suggestive of clinically significant symptoms.

SECONDARY OUTCOMES:
Mini-mental State Examination（MMSE） | 3 months
  The MMSE consists of 2 parts: language (time orientation (5 items), registration and attention) and performance (recall, response to written/verbal commands, sriting ability and reproduction of complex polygons); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
Montreal Cognitive Assessment Scale（MoCA） | 3 months
  The MoCA explores 8 cognitive domains: visuospatial/executive (score range form 0 to 5), naming(0-3), attention (0-5), language (0-3), abstraction(0-2), delayed recall(0-5), and orientation(0-6). The MoCA score was not corrected according to education level as advised by Gagnon and colleagues (2013). Its normal value was≥26 as proposed. A lower score indicates more severe cognitive impairment.
Named test of the Aphasia Battery of Chinese | 3 months
  The Aphasia Battery of Chinese(ABC) was compiled by Surong Gao et al in 1988 in accordance with the basic principles of aphasia inspection.It is mainly based on the Western Aphasia Battery (WAB), which has been developed through exploration and modification in combination with Chese national conditions and clinical experience.The named test is one of the subtest of the ABC.A total score is then calculated of all items which can range from 0 to 82. A higher score is indicative of worse outcome.
Similarity test | 3 months
  The similarity test includes 13 items scored with a range of 0-2. In each item, participants are given two words or concepts and have to describe how they are similar. A lower score indicates more severe abstract verbal reasoning and semantic knowledge impairment.
Symbol Digit modalities test（SDMT） | 3 months
  The Symbol Digit modalities test（SDMT) consists of nine digit-symbol pairs followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the 90 sec is measured.
Verbal fluency test（VFT） | 3 months
  The verbal fluency test is a kind of psychological test in which participants have to produce as many words as possible from a category in a given time (usually 60 seconds). A 60-second limit for responses within each category was allowed. Higher scores represent better performance.
Logical memory test（LMT） | 3 months
  The Logical Memory, subtest of the WMS-R is a standardized assessment of narrative episodic memory. A short story is orally presented, and the examinee is asked to recall the story immediately.
Delayed memory test（DMT） | 3 months
  Approximately 5 and 30 min later of the Logical memory test, recall of the story is again elicited, which is called delayed memory test.
Digit span test（DST） | 3 months
  In digit span test, participants must recall a series of numbers in order. A lower score indicates more severe working memory, attention, encoding and auditory processing impairment.
Ten point clock test | 3 months
  The ten point clock test is a reliable test of cognitive function. A total score is then calculated of all items which can range from 0 to 10. A higher score is indicative of better outcome.
Uniform Parkinson's Disease Rating Scale Ⅲ（UPDRSⅢ） | 3 months
  The motor section of the Unified Parkinson Disease Rating Scale (UPDRSⅢ) is covers the motor evaluation of disability and includes ratings for tremor, slowness (bradykinesia), stiffness (rigidity), and balance; part IV covers a number of treatment complications including ratings of involuntary movements (dyskinesias), painful cramps (dystonia), and irregular medication responses (motor fluctuations). It consists of 27 items, each are scored with a range of 0-4, with total score ranges from 0 to108. A higher score is indicative of more severe motor symptoms.
Modified Hoehn & Yahr scale（H-Y） | 3 months
  The Hoehn&Yahr scale is a commonly used system for describing how the symptoms of Parkinson's disease progress. It was originally published in 1967 in the journal Neurology by Melvin Yahr and Margaret Hoehn and included stages 1 through 5. Since then, a modified Hoehn&Yahr scale was proposed with the addition of stages 1.5 and 2.5 to help describe the intermediate course of the disease. A higher score is indicative of more severe movement impairment.
Time up and go test（TUG test） | 3 months
  The Timed Up and Go Test is well known and widely used where the clinical goal is to get an accurate objective assessment of balance. It measures the time taken by an individual to stand up from a standard arm chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down.
Activity of Daily Living Scale（ADL） | 3 months
  ADL was developed by Lawton and Brody in 1969.It consists of Physical self-maintenance Scale (PSMS) and Instrumental Activities of Daily Living Scale (IADL).It is mainly used to assess the daily life ability of the subjects. The total score below 14 points is indicative normal.More than 16 points is indicative functional decline.The highest score is 56.
Parkinson's Disease Questionnaire（PDQ-39） | 3 months
  The Parkinson's Disease Questionnaire is designed to address aspects of functioning and well-being for those affected by Parkinson's disease. Substantial evidence is available to suggest that the PDQ is reliable, valid, responsive, acceptable and feasible as the tool for the assessment of quality of life in Parkinson's disease patients. There are 39 questions in the long form Parkinson's Disease Questionnaire, with 8 discrete scales:mobility (10 items),activities of daily living (6 items),emotional well-being (6 items),stigma (4 items),social support (3 items),cognitions (4 items),communication (3 items),bodily discomfort (3 items) . Items are scored with a range of 0-4. A total score is then calculated of all items which can range from 0 to 156. A higher score is indicative of worse outcome.
Non-motor symptoms questionnaire(NMS-Q) | 3 months
  The non-motor symptoms (NMS) questionnaire can be given to people affected by Parkinson's in order to aid health and social care professionals to assess their non-motor symptoms.The non-motor symptoms questionnaire is a 30-point, patient-based questionnaire used to determine the non-motor symptoms experienced by the patient during the past month. The points should be totalled to give a score out of 30. A score of under 10 is mild, 10-20 moderate and over 20, severe.
Pittsburgh Sleep Quality Index (PSQI) | 3 months
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. A total score is then calculated of all items which can range from 0 to 21. A higher score is indicative of worse outcome.
Hamilton Anxiety Scale（HAMA） | 3 months
  The Hamilton Anxiety Rating Scale (HAMA) is a designed to assess symptoms of anxiety. Items are scored with a range of 0-4. A total score is then calculated of all items which can range from 0 to 54. A higher score is indicative of more anxiety symptoms, and a lower score post-tx is indicative of better outcome.
Beck Anxiety Inventory（BAI） | 3 months
  The Beck Anxiety Inventory (BAI) is a 21-item self-report questionaire that measures Anxiety symptoms. Each item is scored on a scale of 0-3, and items are summated to yield a total score. A higher score is indicative of greater symptoms of anxiety. Total scores may range between 0 and 63. A score greater than or equal of 8 is suggestive of clinically significant symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Wang, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (10):
- China (10):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Affiliated Union Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brys M, Fox MD, Agarwal S, Biagioni M, Dacpano G, Kumar P, Pirraglia E, Chen R, Wu A, Fernandez H, Wagle Shukla A, Lou JS, Gray Z, Simon DK, Di Rocco A, Pascual-Leone A. Multifocal repetitive TMS for motor and mood symptoms of Parkinson disease: A randomized trial. Neurology. 2016 Nov 1;87(18):1907-1915. doi: 10.1212/WNL.0000000000003279. Epub 2016 Oct 5. PMID 27708129
- [Result] Kojovic M, Kassavetis P, Bologna M, Parees I, Rubio-Agusti I, Berardelli A, Edwards MJ, Rothwell JC, Bhatia KP. Transcranial magnetic stimulation follow-up study in early Parkinson's disease: A decline in compensation with disease progression? Mov Disord. 2015 Jul;30(8):1098-106. doi: 10.1002/mds.26167. Epub 2015 Mar 5. PMID 25753906
- [Result] Dagan M, Herman T, Mirelman A, Giladi N, Hausdorff JM. The role of the prefrontal cortex in freezing of gait in Parkinson's disease: insights from a deep repetitive transcranial magnetic stimulation exploratory study. Exp Brain Res. 2017 Aug;235(8):2463-2472. doi: 10.1007/s00221-017-4981-9. Epub 2017 May 16. PMID 28509934